CLINICAL TRIAL: NCT02956109
Title: Relative Bioavailability Study to Investigate the Pharmacokinetics, Safety and Tolerability of Single Oral Doses of Finerenone 1.25 mg and 5 x 0.25 mg Orodispersible Tablet (Pediatric Formulation) in Comparison to 10 mg Tablet (Adult Formulation) in the Fasting Condition and to Investigate the Effect of a High Fat, High Calorie Meal on 1.25 mg Oro-dispersible Tablet in Healthy Male Subjects in a Randomized, Open-label, Four-fold Crossover Design
Brief Title: Study of Finerenone to Investigate a Paediatric Formulation in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18290; 2016-002895-29 (EudraCT Number)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — finerenone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult formulation: Finerenone tablet_Fasting (Active Comparator): Single oral dose of 10 mg finerenone tablet fasting
  Interventions: Drug: Finerenone (BAY94-8862): 1 0mg tablet
- Pediatric formulation: 5X 0.25 mg Finerenone ODT_Fasting (Experimental): Single oral dose of 5 x 0.25 mg finerenone oro-dispersible tablets fasting
  Interventions: Drug: Finerenone (BAY94-8862): 5 X 0.25 mg oro-dispersible tablets
- Pediatric formulation: 1.25 mg Finerenone ODT_Fasting (Experimental): Single oral dose of 1.25 mg finerenone oro-dispersible tablet fasting
  Interventions: Drug: Finerenone (BAY94-8862): 1.25 mg oro-dispersible tablet
- Pediatric formulation: 1.25 mg Finerenone ODT_Fed (Experimental): Single oral dose of 1.25 mg finerenone oro-dispersible tablet fed; 30 minutes after start of an American breakfast
  Interventions: Drug: Finerenone (BAY94-8862): 1.25 mg oro-dispersible tablet

INTERVENTIONS:
Drug: Finerenone (BAY94-8862): 1 0mg tablet — 10 mg finerenone immediate-release tablet; single dose in the fasting condition
  Arms: Adult formulation: Finerenone tablet_Fasting
Drug: Finerenone (BAY94-8862): 5 X 0.25 mg oro-dispersible tablets — 5 x 0.25 mg (1.25 mg) oro-dispersible tablets; single dose in the fasting condition
  Arms: Pediatric formulation: 5X 0.25 mg Finerenone ODT_Fasting
Drug: Finerenone (BAY94-8862): 1.25 mg oro-dispersible tablet — 1.25 mg finerenone oro-dispersible tablets; single dose in the fasting condition or in the fed condition
  Arms: Pediatric formulation: 1.25 mg Finerenone ODT_Fasting; Pediatric formulation: 1.25 mg Finerenone ODT_Fed

SUMMARY:
Finerenone is developed for the treatment of diabetic kidney disease (adults) and chronic kidney disease (children). The purpose of the proposed trial is to test the pharmacokinetics of a single oral dose of finerenone (1.25 mg tablet and 5 x 0.25 mg tablets) using a novel orodispersible tablet formulation for the treatment of children, in comparison to the adult tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age: 18 to 45 years (inclusive)
* Body mass index (BMI) : ≥ 18 and ≤ 29.9 kg/m²
* Race: White

Exclusion Criteria:

* Subjects with conspicuous findings in medical history and pre-study examination in the opinion of the investigator
* A history of relevant diseases of vital organs, of the central nervous system or other organs
* Known renal or liver insufficiency
* Subjects with diagnosed malignancy, psychiatric disorders, or thyroid disorders (evaluated by medical history, physical examination, clinical symptoms, and assessment of thyroid stimulating hormone at screening)
* Medical disorder that would impair the subject's ability to complete the study in the opinion of the investigator
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Smoking more than 10 cigarettes daily and/ or inability to refrain from smoking on the profile days until 8 h after administration
* Vegetarian or special diets preventing the subjects from eating the standard meals during the study, especially the high-fat high-calorie American breakfast or reluctance to ingest it

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Finerenone area under the plasma concentration vs. time curve (AUC) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5. 3, 4, 6, 8, 12, 15 and 24 hours
Finerenone maximum plasma concentration (Cmax) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5. 3, 4, 6, 8, 12, 15 and 24 hours
Appearance of oro-dispersible tablets assessed by questionnaire | Up to 5 minutes after drug administration
Taste of oro-dispersible tablets assessed by questionnaire | Up to 5 minutes after drug administration
Texture of oro-dispersible tablets assessed by questionnaire | Up to 5 minutes after drug administration
Smell of oro-dispersible tablets assessed by questionnaire | Up to 5 minutes after drug administration
Overall impression of oro-dispersible tablets assessed by questionnaire | Up to 5 minutes after drug administration
Whether oro-dispersible tablets are palatable and swallowable assessed by questionnaire | Up to 5 minutes after drug administration

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany